CLINICAL TRIAL: NCT02649803
Title: Pediatric Asthma Control Under Community Management Model in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ESR-15-10989
Record Dates: First submitted 2016-01-01; First posted 2016-01-07 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
Keywords: pediatric; asthma control; community
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- community hospital (Other): During the study, subjects who diagnosed as asthma according to "Guideline for the diagnosis and optimal management of asthma in children" will be assigned to the nearest community hospital or Shanghai Children's Medical Center, and receive 12 months standard treatment, prescribed by the investigators according to "Guideline for the diagnosis and optimal management of asthma in children". The patient's caregiver will be instructed to install asthma APP at their smart phone to follow up.
  Interventions: Behavioral: asthma APP

INTERVENTIONS:
Behavioral: asthma APP — Subjects diagnosed as pediatric asthma at Shanghai Children's Medical Center will be consecutively screened and eligible patients will be recruited (enrolment visit, V1). The subject will be assigned to the nearest community hospital or Shanghai Children's Medical Center, whichever is nearer to the subject's home, for their future onsite visits (V2-V5). The patient's caregiver will be instructed to install the asthma APP at their smart phone and learn how to use this APP.
  Other Names: study-specified asthma application program

SUMMARY:
The purpose of this study is to learn the pediatric asthma control status under community management model. To learn the differences of pediatric asthma control status when subjects assigned to community hospitals or Shanghai Childrens Medical Centre. To learn the treatment adherence and the frequency of asthma attack under community management model.

DETAILED DESCRIPTION:
Subjects diagnosed as pediatric asthma at Shanghai Children's Medical Center will be consecutively screened and eligible patients will be recruited. For each enrolled patient, basic information as well as baseline medical condition will be collected by the investigators. Asthma medicine will be prescribed by the investigator according to patient's asthma severity and control status. The subject will be assigned to the nearest community hospital or Shanghai Children's Medical Center, whichever is nearer to the subject's home, for their future onsite visits. The patient's caregiver will be instructed to install the study-specified application program (APP) at their smart phone and learn how to use this APP.

During the study, patients will receive 12 months standard treatment, prescribed by the investigators according to "Guideline for the diagnosis and optimal management of asthma in children".

The patients' caregiver will be prompted to fill out an asthma control questionnaire and asthma control test via their smart phone APP every month.

Patients will be requested to visit prearranged community hospitals at month 1, 3, 6, 9 and arrange their last visit back to Shanghai Children's Medical Center at month 12. During each onsite visit, asthma-related information will be collected by the investigators.

Meanwhile, subjects will receive PEF (>5 years old) and FENO tests for evaluation of lung function and inflammation level. After comprehensive assessment of the patient's symptom control, risk factors, occurrence of exacerbations, and practical issues (cost, ability to use the device, and adherence), the investigator will make the decision on whether stepping up or stepping down asthma treatment.

This study ends up without follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Out-patient, female or male, aged less than 18 years old
2. Diagnosed as asthma according to "Guideline for the diagnosis and optimal management of asthma in children"
3. Consent should be obtained by subjects' guardian
4. The subjects or subjects' caregiver must have a smart phone at their disposal

Exclusion Criteria:

1. Presenting with differential diagnosis of asthma such as congenital heart disease, gastro-oesophageal reflux, bronchopulmonary dysplasis, bronchiolitis obliterans, etc.
2. Allergy to any inhaler cortical steroid
3. Subject with other diseases that may interfere the study results judged by the investigators.
4. Participation in any analogous clinical study within 3 months

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 800 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
asthma control questionnaire | 1 year
  The patients' caregiver will be prompted to fill out an asthma control questionnaire via their smart phone APP every month. This questionnaire contains questions regarding renewal of prescription, adherence, control status, asthma attack and health economic information.

SECONDARY OUTCOMES:
asthma control test | 1 year
  caregiver will also be asked to fill out an asthma control test (for patients 12 years or older) , childhood asthma control test (for patients aged 5-12) , or GINA assessment of asthma control in children 5 years and younger.

OTHER OUTCOMES:
FENO tests | 1 year
  Subjects will receive FENO(Fractional exhaled nitric oxide, parts per billion, ppb) tests for evaluation of lung inflammation level.
PEF (>5 years old) | 1 year
  Subjects(older than 5 years) will receive PEF (Peak expiratory flow, L/min) tests for evaluation of lung function.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Yin, PhD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai children's medical center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Zhao L, Zhao D, Chen Z, Li S, Zhang H, Zhang L, Yuan S, Tang M, Wu Y, Zhong W, Xu J, Zhao LX, Liu SY, Hong J, Yin Y. Reliability and validity of the Chinese version of the Test for Respiratory and Asthma Control in Kids (TRACK) in preschool children with asthma: a prospective validation study. BMJ Open. 2019 Aug 26;9(8):e025378. doi: 10.1136/bmjopen-2018-025378. PMID 31455696